CLINICAL TRIAL: NCT06416293
Title: Widening Aims and Giving Patients a Voice for Expanded Structures in Breast Cancer Care Jointly Developed by Patients and Physicians (Wechselseitiger Patienten-Arzt-Austausch in Der Versorgung Bei Brustkrebs Mit Dem Ziel Der Gemeinsamen Erarbeitung Neuer Patienten-orientierter Strukturen)
Brief Title: Widening Aims and Giving Patients a Voice for Expanded Structures in Breast Cancer Care Jointly Developed by Patients and Physicians
Acronym: WAVES
Status: Recruiting | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Collaborators: Wuerzburg University Hospital (Other); Technical University of Munich (Other); LMU Klinikum (Other); University Hospital Regensburg (Other); University Hospital Erlangen (Other); Bavarian Cancer Research Center (BZKF) (Unknown)
Responsible Party: Principal Investigator, Nina Ditsch, Head of Breast Centre University Hospital Augsburg, Principal Investigator, Clinical Professor, University Hospital Augsburg
Other Study IDs: 2.0
Record Dates: First submitted 2024-04-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Communication; patient-physician-relationship; questionnaire
MeSH Terms: conditions — Breast Neoplasms; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BC Patients: Patients with diagnosis of breast cancer or DCIS
  Interventions: Other: Questionnaire patients
- Physicians: Physicians treating patients with breast cancer
  Interventions: Other: Questionnaire physicians

INTERVENTIONS:
Other: Questionnaire patients — Completion of a two-part questionnaire with a special focus on communication around the breast cancer diagnosis. Tumor stage and therapies received are also surveyed. The questionnaire can be answered online via a secure tool (REDCap) or in paper form.
  Groups: BC Patients
Other: Questionnaire physicians — Completion of a questionnaire with a special focus on communication around the breast cancer diagnosis
  Groups: Physicians

SUMMARY:
The aim of this BZKF project is to record the current care structure for breast cancer patients in order to use this as a basis for developing possible future models for improvement. The active involvement of representatives of regional and national patient organizations in the creation of a patient-based and patient-oriented survey ensures that the needs of patients are the focus. In addition to and in contrast to other projects, relevant questions are explicitly addressed not only to patients but also to physicians in order to identify and specify the interfaces between patient wishes/suggestions and to develop clinical consequences for care.

The first objective is to survey the "current situation" by recording the current care structure for breast cancer. The focus is on the survey of both groups on patient-physician communication, time management and coping strategies.

By planning the future harmonization of national data structures, the basis is created for the long-term goal of an improved "target", a concept developed jointly by physicians and patients for an improved communication and care structure that focuses on the patient.

ELIGIBILITY:
Inclusion Criteria (patients):

* Breast cancer or DCIS
* women and men aged 18 years and older

Exclusion Criteria (patients):

* women and men < 18 years
* no histologically confirmed breast cancer or DCIS diagnosis

Inclusion Criteria (physicians):

- Treatment of breast cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women and men aged 18 years and older with breast cancer. Physicians treating breast cancer patients.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Current state of care - patient view | through study completion, an average of 3 years
  The primary aim of the questionnaire is to record the current reality of care for breast cancer patients with a focus on communication.

SECONDARY OUTCOMES:
Current state of care - physician view | through study completion, an average of 3 years
  Secondarily, a comparison will be made with the physicians assessment of the same topics

CONTACTS AND LOCATIONS:
Overall Officials: Nina Ditsch, Prof., Principal Investigator — University Hospital Augsburg
Locations (1):
- University Hospital Augsburg, Department of Gynecology and Obstetrics, Augsburg, Bavaria, Germany